CLINICAL TRIAL: NCT06513598
Title: New Studies of the Pathogenesis of Postoperative Infections and Development of Biomarkers for Early Diagnosis of Postoperative Complications
Brief Title: Pathogenesis of Postoperative Infections and Biomarkers for Early Diagnosis of it
Status: Recruiting | Type: Observational
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Augustinas Bausys, Principal Investigator, National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos
Other Study IDs: 1v3
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Complication of Surgical Procedure; Infections
Keywords: microbiota; surgical oncology; gastrointestinal cancer; postoperative complications; biomarkers
MeSH Terms: conditions — Infections; Gastrointestinal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1) Stool samples; 2) oral cavity swabs; 3) blood 4) samples from infection sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Major visceral surgery for gastrointestinal cancer — This is a longitudinal observational study of the patients undergoing major visceral surgery for gastrointestinal cancer. Biological samples will be collected to compare gastrointestinal and infection site metastases and develop biomarkers for postoperative infections.

SUMMARY:
Infections remain a prevalent complication after major abdominal surgery. The common belief that most surgical site infections (SSIs) following elective surgery with modern antiseptic techniques are due to intraoperative contamination is still not confirmed. Therefore, alternative mechanisms for SSI development, such as the Trojan Horse theory-which suggests that pathogens from distant sites like the gastrointestinal tract may cause postoperative infections-should be explored. This study aims to analyze the preoperative microbiome of surgical patients' gut and oral cavities and assess whether microorganisms found there are present at the infection site. Additionally, this study will investigate a panel of biomarkers for predicting postoperative infections.

DETAILED DESCRIPTION:
Infections remain a significant concern following major abdominal surgery. The prevailing notion that most surgical site infections (SSIs) after elective surgery with modern antiseptic techniques are solely caused by intraoperative contamination remains unconfirmed. Therefore, alternative mechanisms for SSI development, such as the Trojan Horse theory-which suggests that pathogens from distant sites like the gastrointestinal tract may contribute to postoperative infections-require thorough investigation. This longitudinal observational study aims to either support or challenge the Trojan Horse theory.

This study will enroll patients undergoing major abdominal surgery for confirmed or suspected cancer. Biological samples from stool, the oral cavity, and infection sites will be collected for sequencing and microbiome analysis to evaluate the presence of pathogens potentially responsible for postoperative infections originating from the gastrointestinal tract. Additionally, blood samples will be collected to identify predictive biomarkers associated with the development of postoperative infections.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is scheduled to undergo a major resection-type abdominal surgery due to cancer of the esophagus, stomach, pancreas, liver, bile ducts, colon or rectum.
2. Patient is willing to participate.
3. Age ≥ 18 years.

Exclusion Criteria:

1. Pregnancy.
2. Previous surgical resection of the digestive tract, excluding appendectomy and/or cholecystectomy.
3. Anticipated operation with preventive ileostomy.
4. The operation is planned to be performed as a matter of urgency.
5. Antibiotic therapy ≤1 month. before surgery.
6. Chronic inflammatory bowel disease (non-specific ulcerative colitis, Crohn's disease) or radiation or other colitis of origin.
7. During the last year, the patient suffered from Cl. difficile colitis or was Cl. difficile carrier, had salmonellosis or others intestinal infections.
8. During the last year, the patient used (> 3 months) pre-/pro-/(syn)biotics.
9. During the last year, the patient has been taking proton pump inhibitors continuously (> 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo major abdominal surgery due to the cancer of the esophagus, stomach, pancreas, liver, bile ducts, colon, or rectum due to cancer will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
The similarity in composition between the infection site microbiome and the gut/oral microbiome. | 0 to 30 days

SECONDARY OUTCOMES:
Incidence of postoperative infections after major abdominal surgery for gastrointestinal cancer. | 0 to 30 days
  Infections diagnosed within 30 days after surgery
Incidence of surgical site infections after major abdominal surgery for gastrointestinal cancer. | 0 to 30 days
  A surgical site infection (SSI) is an infection in the part of the body where a surgery took place.
Major abdominal resection impact on gut microbiome composition. | 0 to 30 days
  Baseline and POD6 gut microbiome composition will be compared.
Gut microbiome-based biomarkers for postoperative infections. | 0 to 30 days
Intestinal wall permeability and local inflammatory markers (LBP, I-FABP, sCD14, etc.) will be evaluated as a potential biomarkers for postoperative infections. | 0 to 30 days
  Intestinal wall permeability and local inflammatory markers (LBP, I-FABP, sCD14, etc.) on PODs2, 3 and 4 will be evaluated as potential biomarkers for postoperative infections.
Inflammatory cytokines (IL4; IL2; IP10; IL1β; TNFα; etc.) and pro-inflamatory microRNAs (miRNA-21, miRNA-155, etc.) will be evaluated as a potential biomarkers for postoperative infections. | 0 to 30 days
  Inflammatory cytokines (IL4; IL2; IP10; IL1β; TNFα; etc.) and pro-inflamatory microRNAs (miRNA-21, miRNA-155, etc.) on PODs2, 3 and 4 will be evaluated as potential biomarkers for postoperative infections.
The proportion of patients developing wound infections among those with positive and negative wound cultures at the conclusion of surgery. | 0 to 30 days
  Wound swabs will be taken for culture at the end of surgery before closing skin. Proportion of patients developing wound infection among patients with positive and negative culture will be determined.

CONTACTS AND LOCATIONS:
Locations (2):
- Lithuania (2):
  - National Cancer Institute, Vilnius
  - Vilnius University hospital Santaros Klinikos, Vilnius

IPD SHARING:
Plan to Share IPD: No